CLINICAL TRIAL: NCT02303314
Title: Efficacy of Oral Trigonella Foenum-graecum Seed Extract Vs Placebo in Treatment of None Alcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Hossein Babaei, Students of Medicine, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P-9362-6352; IRCT2013102015083N1 (Registry Identifier: Iranian Registry of Clinical Trials); CT-P-9362-6352 (Other: Shirazums)
Record Dates: First submitted 2014-11-21; First posted 2014-11-27 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug: Trigonella Foenum-graecum (Other): in this group patients use Trigonella Foenum-graecum seed extract twice daily.
  Interventions: Drug: Trigonella Foenum-graecum Seed Extract
- Drug: Placebo (Other): in this group patients use placebo twice daily.
  Interventions: Drug: Drug: Placebo

INTERVENTIONS:
Drug: Trigonella Foenum-graecum Seed Extract
  Arms: Drug: Trigonella Foenum-graecum
Drug: Drug: Placebo
  Arms: Drug: Placebo

SUMMARY:
This study design to examine performance of trigonella foenum-graecum (TFG) in treatment of non-alcoholic fatty liver disease. Base on inclusion and exclusion criteria, 50 patients select and then randomize into intervention and control groups. Two group use capsules which contain TFG or placebo, respectively.

DETAILED DESCRIPTION:
This study design to examine performance of trigonella foenum-graecum in treatment of non-alcoholic fatty liver disease. Patients 18-70 year old with the levels of ALT and AST greater than 1.5 and less than 10 times normal level, and ultrasound evidence confirm fatty liver disease include in study. Patients with alcohol consumption, other liver disease and taking medications that cause liver injury, exclude. Base on inclusion and exclusion criteria, 50 patients select and then randomize into intervention and control groups. Control group, in addition to diet and exercise recommendations take placebo capsules for 3 months. Intervention group, in addition to diet and exercise recommendations, use capsules containing hydro-alcoholic extract of fenugreek 1g/d for 3 months. At baseline and 6 and 12 weeks after intervention, the investigators measure FBS, insulin, insulin resistance, Albumin, Aspartate transaminase, Alanine Aminotransferase, Alkaline phosphatase, Total bilirubin, Direct bilirubin, HbA1c, total cholesterol, LDL, HDL, TG, High sensitivity C reactive protein and Creatinine. At baseline and 12 weeks after intervention fibroscan perform to evaluate the amount of fat in liver. In order to decrease bias, patient, physician who performs fibroscan and the person analyzing the data are blind to group drugs.

ELIGIBILITY:
Inclusion criteria:

* The level of ALT and AST greater than 1.5 and less than 10 times normal level
* Ultrasound evidence confirm fatty liver disease; age between 18-70 years old
* Negative pregnancy test for women in reproductive age (up to two weeks prior to the study)
* Negative for hepatitis B and C
* BMI: 18.5 to 40
* Sign the consent form.

Exclusion criteria:

* History of more than one unit of alcohol consumption (one value for the Spirits (vodka; whiskey)
* Wine and Beer are respectively 30-45 cc; 120-150 cc and 360 cc.)
* Fatty liver controller medications
* Glucose lowering drugs
* Cholesterol lowering drugs
* Hypotensive drugs
* Consumption of vitamin E
* Taking coenzyme Q10
* Administration of corticosteroids & glucocorticoids
* Thyroxin administration
* Administration of drugs that cause fatty liver
* Diabetes (type 1 and 2)
* History of cancer in the past
* Hepatocellular carcinoma
* Renal failure (creatinine> 1.5 x ULN)
* Chronic pancreatitis
* Cirrhosis
* Uncontrolled hypertension (above 180 mm Hg systolic blood pressure); heart disease
* Autoimmune hepatitis
* Primary biliary cirrhosis
* Primary sclerosing cholangitis (alkaline phosphatase levels greater than 3 times normal)
* Wilson's disease
* Alpha-1 antitrypsin deficiency and coronary artery disease
* Symptoms of hypothyroidism
* Hyperthyroidism
* Disorders of the hypothalamic - pituitary
* Liver transplantation
* Pregnant or lactating women
* Those who cannot use contraceptives.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-11; Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Liver stiffness change | At baseline and 12 weeks after intervention
  Assessment by Fibroscan

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Alireza Taghavi, Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran